CLINICAL TRIAL: NCT03927001
Title: Prospective, Open-Label, Multi-Center Single-Arm Trial Designed to Assess the Safety, Performance and Efficacy of the NeVa Stent Retriever in the Treatment of Large Vessel Occlusion Strokes
Brief Title: The Vesalio NeVa Stent Retriever Study for Treatment of Large Vessel Occlusion Strokes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vesalio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-006 / G
Record Dates: First submitted 2019-04-18; First posted 2019-04-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Intervention (Other): NeVa Stent Retrievers
  Interventions: Device: NeVa Stent Retrievers

INTERVENTIONS:
Device: NeVa Stent Retrievers — mechanical neurothrombectomy

SUMMARY:
A prospective, open label, single-arm 90-day study designed to assess the safety, performance and efficacy of thrombus removal in subjects presenting with acute ischemic stroke with the NeVa stent retrievers.

DETAILED DESCRIPTION:
This is a prospective, open label, multi-center, single-arm trial designed to assess the safety, performance and efficacy of the NeVa stent retriever in the treatment of large vessel occlusion strokes. Up to 150 subjects at up 20 sites will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical signs and symptoms consistent with the diagnosis of an acute ischemic stroke, and subject belongs to one of the following subgroups:

   1.1. Subject has failed IV t-PA therapy

   1.2. Subject is contraindicated for IV t-PA administration

   1.3. IV-tPA given within 3 hours of symptom onset
2. Age ≥18 and less than equal to 85
3. NIHSS score ≥ 8 and ≤ 25
4. Prestroke mRS score of ≤ 1
5. Intracranial arterial occlusion of the distal intracranial carotid artery or middle cerebral artery (M1/M2), anterior cerebral artery (ACA), posterior cerebral artery (PCA), basilar artery, or vertebral artery demonstrated with DSA.
6. Thrombectomy procedure can be initiated within 8 hours from symptom onset (defined as time last known well [TLKW]) and at least one NeVa pass occurring within 8 hours
7. Imaging Inclusion Criteria:

   7.1. Non-Contrast CT Selection (if CT Perfusion or MRI not utilized): ASPECTS 6-10 , or

   7.2. CT Perfusion core ≤50 cc, or

   7.3. MRI DWI core ≤50 cc
8. Subject or (legal) representative or independent physician (if approved by site's regional ethics committee, see site's informed consent form) is able and willing to give informed consent prior to the interventions.

Exclusion Criteria:

1. Pre-existing medical neurological or psychiatric disease that would confound the neurological or functional evaluations, e.g. dementia with prescribed anti-cholinesterase inhibitor (e.g. Aricept).
2. Cardiopulmonary resuscitation, significant cardiac arrhythmia, evidence of ongoing myocardial infarction, concern for pre-treatment pulmonary aspiration.
3. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
4. Cerebral vasculitis
5. History of severe allergy to contrast medium.
6. Known allergy to NeVa materials (nitinol, stainless steel);
7. Suspicion of aortic dissection, septic embolus, or bacterial endocarditis
8. Systemic infection
9. Significant mass effect with midline shift
10. Evidence of intracranial tumor (except small meningioma [≤ 3cm])
11. Any CT or MRI evidence of acute hemorrhage products on presentation
12. Inability to deploy NeVA device for at least one pass for any other reason
13. Life expectancy less than 6 months
14. Any other condition that, in the opinion of the investigator, precludes an endovascular procedure or poses a significant hazard to the subject if an endovascular procedure was performed.
15. Active malignancy
16. Stenosis or occlusion in a proximal vessel requiring treatment or preventing access to the thrombus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Recanalization rate of the occluded target vessel | post-procedure day 0
  Recanalization rate of the occluded target vessel (defined by an eTICI score ≥ 2b) following three or less passes using the NeVa device(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Vall d'Hebron, Barcelona, Spain